CLINICAL TRIAL: NCT05716269
Title: Evaluation of Visual Outcomes and Patient Satisfactory After PanOptix Implantation in Hyperopic Cataract Patients: a Prospective, Cohort Study
Brief Title: Visual Outcomes and Patient Satisfactory After PanOptix Implantation in Hyperopic Cataract Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Tianjin Eye Hospital (Other)
Responsible Party: Principal Investigator, Hong Qi, Professor, Peking University Third Hospital
Other Study IDs: 2022756
Record Dates: First submitted 2023-01-22; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cataract; Hyperopia
MeSH Terms: conditions — Cataract; Hyperopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate visual outcomes and patient satisfactory after PanOptix implantation in hyperopic cataract patients

DETAILED DESCRIPTION:
Patients with axial length ≤22.5mm will be recruited. The subjects will undergo bilateral uneventful phacoemulsification and implantation of PanOptix. Visual quality and patients satisfactory will be assessed three months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* age-related cataract patients

  * Eye axis length ≤22.5mm and refraction ≥ +0.5D
  * Predicted postoperative corneal astigmatism ≤0.75D
  * mesopic pupil size between 3.0mm to 5.5 mm
  * Preoperative angle kappa ≤ 0.5 mm
  * Preoperative corneal spherical aberration <0.5μm, high order aberration <0.5μm

Exclusion Criteria:

* In the presence of other ocular diseases that may affect the stability of the lens capsule (pseudoexfoliation syndrome, glaucoma, traumatic cataract, Marfan syndrome, etc.)
* Pupil abnormality (non-reactive pupil, tonic pupils, abnormally shaped pupils, etc.)
* History of any clinically significant retinal pathology or ocular diagnosis (e.g. diabetic retinopathy, ischemic diseases, macular degeneration, retinal detachment, optic neuropathy optic nerve atrophy, amblyopia, strabismus, microphthalmos, aniridia, epiretinal membrane etc.) in the study eyes that could alter or limit final postoperative visual prognosis
* Patients with history of ocular trauma or prior ocular surgery including refractive procedures
* Preoperative visual acuity of worse than 0.2 logMAR in any eye.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hyperopic cataract patients receiving bilateral uneventful phacoemulsification and implantation of PanOptix.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Best corrected distance visual acuity of the operated eye | 3 months postoperatively
  Best corrected distance visual acuity (BCDVA) of the operated eye will be measured.

SECONDARY OUTCOMES:
Uncorrected distance visual acuity (UCVA) | 3 months postoperatively
  Uncorrected distance visual acuity (UCVA) of the operated eye will be measured at 5m.
Uncorrected intermediate visual acuity | 3 months postoperatively
  Uncorrected intermediate visual acuity of the operated eye will be measured at 60cm and 80cm respectively.
Uncorrected near visual acuity | 3 months postoperatively
  Uncorrected near visual acuity of the operated eye will be measured at 40cm.
Best corrected intermediate visual acuity | 3 months postoperatively
  Best corrected intermediate visual acuity of the operated eye will be measured at 60cm and 80cm respectively.
Best corrected near visual acuity | 3 months postoperatively
  Best corrected near visual acuity of the operated eye will be measured at 40cm.
Manifest refraction spherical equivalent | 3 months postoperatively
  Manifest refraction spherical equivalent of the operated eye will be measured
Visual disturbance, spectacle independence and patient satisfaction | 3 months postoperatively
  A questionnaire including visual disturbance, spectacle independence and patient satisfaction will be distributed to subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, MD, PhD, Principal Investigator — Peking University Third Hospital